CLINICAL TRIAL: NCT03659032
Title: Efficacy of Pediatric Manual Therapy in the Positional Plagiocephaly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Iñaki Pastor Pons, Researcher at PhD School, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PMT1
Record Dates: First submitted 2018-09-01; First posted 2018-09-06 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Plagiocephaly; Plagiocephaly, Nonsynostotic; Plagiocephaly, Positional
Keywords: Manual Therapy; Cranial assymmetry; Cranial deformation; Physical Therapy
MeSH Terms: conditions — Plagiocephaly; Plagiocephaly, Nonsynostotic | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Investigator, Outcomes Assessor
Masking Description: The assessors who receive participants and do the measurement are masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pediatric Manual Therapy Group (Experimental): 10 sessions of Pediatric Manual Therapy, once a week. Soft cervical mobilisation, myofascial induction and cranial techniques will be administered. Educational physiotherapy consists in "tummy time" stimulation, visual and kinaesthetic stimulation on the non preferential head position and counter position will be also administered.
  Interventions: Procedure: Pediatric Manual Therapy
- Control Group (Active Comparator): Only Educational Physical Therapy consists in "tummy time" stimulation, visual and kinaesthetic stimulation on the non preferential head position and counter position will be administered.
  Interventions: Procedure: Educational Physical Therapy

INTERVENTIONS:
Procedure: Pediatric Manual Therapy
  Other Names: Manual Therapy; Manual Physical Therapy
  Arms: Pediatric Manual Therapy Group
Procedure: Educational Physical Therapy
  Other Names: Pediatric Physical Therapy
  Arms: Control Group

SUMMARY:
This study evaluates the efficacy of Pediatric Manual Therapy in the treatment of positional plagiocephaly in infants. 40 participants will receive a protocol of Pediatric Manual Therapy and educational physiotherapy in combination, while the other 20 will receive only educational physiotherapy

DETAILED DESCRIPTION:
The Manual Therapy has shown efficacy in different pathologies in the adult but it is not know its utility in infants and children population, nor in specific pathologies as non synostotic plagiocephaly.

In the conservative treatment of plagiocephaly the educational physiotherapy and the helmet therapy have the better level of evidence among other treatments.

A protocol of ten sessions of Pediatric Manual Therapy will be applied to infants with positional plagiocephaly in combination with educational physiotherapy. The protocol consists in soft cervical mobilisation, myofascial induction and the application of some pressures to the cranial bones to improve the asymmetry of the head. Educational therapy which consists in more "tummy time" stimulation, stimulation to the non preference position of the head and counter positioning.

The control group will receive only Educational therapy.

ELIGIBILITY:
Inclusion Criteria:

* Sign of positional plagiocephaly
* Infants below 6 moths age

Exclusion Criteria:

* No neurological disorders
* No infectious diseases
* No respiratory diseases
* No other treatments

Max Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Right Oblique Cranial Vault Diameter | 10 weeks
  Measured with caliper, is the distance from left external part of the orbit to the right lambdoid suture at the horizontal plane
Left Oblique Cranial Vault Diameter | 10 weeks
  Measured with caliper, is the distance from right external part of the orbit to the left lambdoid suture at the horizontal plane

SECONDARY OUTCOMES:
Cranial length | 10 weeks
  Measured with calliper, is the distance from most anterior point in the frontal bone in the middle line to the most posterior point in the cranial vault on the horizontal plane in the middle line
Cranial wide | 10 weeks
  Measured with calliper, is the distance between the two more lateral points in the vault, usually in the temporal or parietal bone.
Cranial circumference | 10 weeks
  Measured in cm with a measuring tape.

CONTACTS AND LOCATIONS:
Overall Officials: Orosia Lucha, Study Director — Universidad de Zaragoza
Locations (1):
- Instituto deTerapias Integrativas, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Billi M, Greco A, Colonneli P, Volpi G, Valente D, Galeoto G. The functional manual therapy intervention in infants with non-synostotic plagiocephaly: a pilot study. Minerva Pediatr (Torino). 2022 Jun;74(3):294-300. doi: 10.23736/S2724-5276.17.04838-1. Epub 2017 Oct 25. PMID 29072040
- [Background] Cabrera-Martos I, Valenza MC, Valenza-Demet G, Benitez-Feliponi A, Robles-Vizcaino C, Ruiz-Extremera A. Effects of manual therapy on treatment duration and motor development in infants with severe nonsynostotic plagiocephaly: a randomised controlled pilot study. Childs Nerv Syst. 2016 Nov;32(11):2211-2217. doi: 10.1007/s00381-016-3200-5. Epub 2016 Jul 27. PMID 27465676
- [Background] Bagagiolo D, Didio A, Sbarbaro M, Priolo CG, Borro T, Farina D. Osteopathic Manipulative Treatment in Pediatric and Neonatal Patients and Disorders: Clinical Considerations and Updated Review of the Existing Literature. Am J Perinatol. 2016 Sep;33(11):1050-4. doi: 10.1055/s-0036-1586113. Epub 2016 Sep 7. PMID 27603533
- [Background] Xia JJ, Kennedy KA, Teichgraeber JF, Wu KQ, Baumgartner JB, Gateno J. Nonsurgical treatment of deformational plagiocephaly: a systematic review. Arch Pediatr Adolesc Med. 2008 Aug;162(8):719-27. doi: 10.1001/archpedi.162.8.719. PMID 18678803
- [Background] Ballardini E, Sisti M, Basaglia N, Benedetto M, Baldan A, Borgna-Pignatti C, Garani G. Prevalence and characteristics of positional plagiocephaly in healthy full-term infants at 8-12 weeks of life. Eur J Pediatr. 2018 Oct;177(10):1547-1554. doi: 10.1007/s00431-018-3212-0. Epub 2018 Jul 20. PMID 30030600
- [Background] Kunz F, Schweitzer T, Grosse S, Wassmuth N, Stellzig-Eisenhauer A, Bohm H, Meyer-Marcotty P, Linz C. Head orthosis therapy in positional plagiocephaly: longitudinal 3D-investigation of long-term outcomes, compared with untreated infants and with a control group. Eur J Orthod. 2019 Jan 23;41(1):29-37. doi: 10.1093/ejo/cjy012. PMID 29617743
- [Background] Ditthakasem K, Kolar JC. Deformational Plagiocephaly: A Review. Pediatr Nurs. 2017 Mar-Apr;43(2):59-64. PMID 29394478
- [Background] Williams E. Preventing "Flat-headed" Babies: A Commentary on "Impact of Parent Practices of Infant Positioning on Head Orientation Profile and Development of Positional Plagiocephaly in Healthy Term Infants". Phys Occup Ther Pediatr. 2018 Feb;38(1):15-17. doi: 10.1080/01942638.2018.1405661. No abstract available. PMID 29372872
- [Background] Nahles S, Klein M, Yacoub A, Neyer J. Evaluation of positional plagiocephaly: Conventional anthropometric measurement versus laser scanning method. J Craniomaxillofac Surg. 2018 Jan;46(1):11-21. doi: 10.1016/j.jcms.2017.10.010. Epub 2017 Oct 16. PMID 29137851
- [Background] Lam S, Luerssen TG, Hadley C, Daniels B, Strickland BA, Brookshier J, Pan IW. The health belief model and factors associated with adherence to treatment recommendations for positional plagiocephaly. J Neurosurg Pediatr. 2017 Mar;19(3):282-288. doi: 10.3171/2016.9.PEDS16278. Epub 2017 Jan 13. PMID 28084919
- [Background] van Vlimmeren LA, Engelbert RH, Pelsma M, Groenewoud HM, Boere-Boonekamp MM, der Sanden MW. The course of skull deformation from birth to 5 years of age: a prospective cohort study. Eur J Pediatr. 2017 Jan;176(1):11-21. doi: 10.1007/s00431-016-2800-0. Epub 2016 Nov 4. PMID 27815732
- [Background] Aarnivala H, Vuollo V, Harila V, Heikkinen T, Pirttiniemi P, Valkama AM. Preventing deformational plagiocephaly through parent guidance: a randomized, controlled trial. Eur J Pediatr. 2015 Sep;174(9):1197-208. doi: 10.1007/s00431-015-2520-x. Epub 2015 Apr 1. PMID 25823758
- [Background] De Bock F, Braun V, Renz-Polster H. Deformational plagiocephaly in normal infants: a systematic review of causes and hypotheses. Arch Dis Child. 2017 Jun;102(6):535-542. doi: 10.1136/archdischild-2016-312018. Epub 2017 Jan 19. PMID 28104626
- [Derived] Pastor-Pons I, Lucha-Lopez MO, Barrau-Lalmolda M, Rodes-Pastor I, Rodriguez-Fernandez AL, Hidalgo-Garcia C, Tricas-Moreno JM. Efficacy of pediatric integrative manual therapy in positional plagiocephaly: a randomized controlled trial. Ital J Pediatr. 2021 Jun 5;47(1):132. doi: 10.1186/s13052-021-01079-4. PMID 34090515
- [Derived] Pastor-Pons I, Hidalgo-Garcia C, Lucha-Lopez MO, Barrau-Lalmolda M, Rodes-Pastor I, Rodriguez-Fernandez AL, Tricas-Moreno JM. Effectiveness of pediatric integrative manual therapy in cervical movement limitation in infants with positional plagiocephaly: a randomized controlled trial. Ital J Pediatr. 2021 Feb 25;47(1):41. doi: 10.1186/s13052-021-00995-9. PMID 33632268

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-01-09): https://cdn.clinicaltrials.gov/large-docs/32/NCT03659032/SAP_002.pdf
  • Informed Consent Form (2018-01-09): https://cdn.clinicaltrials.gov/large-docs/32/NCT03659032/ICF_003.pdf